CLINICAL TRIAL: NCT01496846
Title: Articaine Versus Lidocaine Supplemental Infiltration Efficacy in Irreversible Pulpitis Mandibular Molars After Failed Inferior Alveolar Nerve Block
Brief Title: Efficacy Study of Articaine Versus Lidocaine as Supplemental Infiltration in Inflamed Molars
Acronym: ARTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Dentsply International (Industry)
Responsible Party: Principal Investigator, Mathilde Peters, DMD, PhD, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PG#N014189; HUM00049692 (Other: U-Michigan); HUM00088384 (Other: U-Michigan)
Record Dates: First submitted 2011-12-09; First posted 2011-12-21 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-09

CONDITIONS: Irreversible Pulpitis
Keywords: Articaine; Lidocaine; Anesthesia, Local; Endodontics; Molar; Dental Pulp Diseases
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Carticaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IANB Articaine (Active Comparator): IANB Articaine: Inferior alveolar nerve block (IANB) anesthesia with articaine local anesthetic.
  Interventions: Drug: IANB Articaine
- SUP Articaine (Active Comparator): SUP Articaine: Supplemental buccal anesthesia (SUP) with articaine local anesthetic after unsuccessful IANB.
  Interventions: Drug: IANB Articaine; Drug: SUP Articaine
- SUP Lidocaine (Active Comparator): SUP Lidocaine: Supplemental buccal anesthesia (SUP) with lidocaine local anesthetic after unsuccessful IANB.
  Interventions: Drug: IANB Articaine; Drug: SUP Lidocaine

INTERVENTIONS:
Drug: IANB Articaine — IANB anesthesia given with 1.7cc of 4% articaine, 1:100,000 epinephrine.
  Other Names: Articadent (Dentsply Pharmaceutical)
Drug: SUP Articaine — After unsuccessful IANB with articaine, proceed to give 1.7cc of 4% articaine with 1:100,000 epinephrine in buccal mucosa as a supplemental infiltration injection (SUP).
  Other Names: Articadent (Dentsply Pharmaceutical)
  Arms: SUP Articaine
Drug: SUP Lidocaine — After unsuccessful IANB with articaine, proceed to give 1.7cc of 2% lidocaine with 1:100,000 epinephrine in buccal mucosa as a supplemental infiltration injection (SUP).
  Other Names: Generic lidocaine (Henry Schein Inc)
  Arms: SUP Lidocaine

SUMMARY:
The purpose of this trial is to study the ability of a frequently used dental anesthetic (articaine) to achieve complete numbness of a diseased tooth with the most commonly used injection technique in the lower jaw (inferior alveolar nerve block: IANB). If this technique fails, a commonly used supplemental (SUP) technique with one of two possible dental anesthetics (lidocaine or articaine) will be given to evaluate the success/failure of complete numbness between the two anesthetics.

Standardized administration of anesthesia is provided by controlled delivery using Midwest Comfort Control Syringe.

The investigators hypothesize that supplemental infiltration anesthesia with articaine will give the same success rate as lidocaine in achieving complete pulpal anesthesia in mandibular molars with irreversible pulpits.

This study consisted of two periods of patient enrollment, treatment and data collection: Part I: 101 subjects; Part II: 100 subjects.

DETAILED DESCRIPTION:
The goal of the study is to achieve complete pulpal anesthesia in irreversible pulpitis mandibular molars, either by IANB administration of 4% articaine with 1:100,000 epinephrine (NDA 022466), or in case the IANB appeared to be clinically unsuccessful by supplemental infiltration of either articaine or lidocaine.

The proposed randomized controlled trial (RCT) aims to answer the following questions:

1. What is the success rate of an IANB with articaine using a conventional IANB technique and standardized speed of administration?
2. Is there a difference in complete pulpal anesthetic efficacy using supplemental infiltration with either articaine or lidocaine after an unsuccessful articaine IANB?
3. Is there a difference in first or second molars in achieving complete pulpal anesthesia using supplemental infiltration with either articaine or lidocaine?

This study will combine the data from HUM00049692- Articaine Efficacy in Inflamed Molars to create a larger sample size, giving a total sample size of approximately 200 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* irreversible pulpitis in mandibular molar

Exclusion Criteria:

* below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2011-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde C Peters, DMD, PhD, Study Chair — University of Michigan; Tatiana Botero, DDS, MS, Study Director — University of Michigan
Locations (1):
- University of Michigan, School of Dentistry Clinics, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brandt RG, Anderson PF, McDonald NJ, Sohn W, Peters MC. The pulpal anesthetic efficacy of articaine versus lidocaine in dentistry: a meta-analysis. J Am Dent Assoc. 2011 May;142(5):493-504. doi: 10.14219/jada.archive.2011.0219. PMID 21531931
- [Result] Rogers BS, McDonald NJ, Gardner R, Botero T, Shlafer M, Peters MC. Anesthetic Efficacy of Articaine vs Lidocaine as Supplemental Infiltration after Unsuccessful IANB of Irreversible Pulpitis Mandibular Molars. AAE Annual Meeting. Honolulu, Hawaii, April 2013.
- [Result] Rogers BS, Botero TM, McDonald NJ, Gardner RJ, Peters MC. Efficacy of articaine versus lidocaine as a supplemental buccal infiltration in mandibular molars with irreversible pulpitis: a prospective, randomized, double-blind study. J Endod. 2014 Jun;40(6):753-8. doi: 10.1016/j.joen.2013.12.022. Epub 2014 Feb 8. PMID 24862701
- [Result] Shapiro MR, McDonald NJ, Gardner RJ, Peters MC, Botero TM. Efficacy of Articaine versus Lidocaine in Supplemental Infiltration for Mandibular First versus Second Molars with Irreversible Pulpitis: A Prospective, Randomized, Double-blind Clinical Trial. J Endod. 2018 Apr;44(4):523-528. doi: 10.1016/j.joen.2017.10.003. Epub 2018 Feb 1. PMID 29397214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol enrollment: 201 subjects with 1 study tooth.
Pre-assignment Details: All enrolled study participants (N=201) initially received an Articaine inferior alveolar nerve block (IANB).
  If unsuccessful (N=149), this was followed by a supplemental dose (SUP) of either Articaine or Lidocaine.
  Fifty-two subjects were excluded prior to assignment to groups due to inadequate lip numbness (N=2) or successful IANB (N=50).
Groups:
- IANB Articaine Only - 1st Molar: IANB anesthesia with articaine local anesthetic provided to 1st Molar.
- IANB Articaine Only - 2nd Molar: IANB anesthesia with articaine local anesthetic provided to 2nd Molar.
- IANB Articaine and SUP Articaine - 1st Molar: Supplemental buccal anesthesia (SUP) with articaine local anesthetic provided to 1st Molar after unsuccessful IANB.
- IANB Articaine and SUP Articaine - 2nd Molar: Supplemental buccal anesthesia (SUP) with articaine local anesthetic provided to 2nd Molar after unsuccessful IANB.
- IANB Articaine and SUP Lidocaine - 1st Molar: Supplemental buccal anesthesia (SUP) with lidocaine local anesthetic provided to 1st Molar after unsuccessful IANB.
- IANB Articaine and SUP Lidocaine - 2nd Molar: Supplemental buccal anesthesia (SUP) with lidocaine local anesthetic provided to 2nd Molar after unsuccessful IANB.
Period: IANB Articaine (All Participants)
Arm/Group | IANB Articaine Only - 1st Molar | IANB Articaine Only - 2nd Molar | IANB Articaine and SUP Articaine - 1st Molar | IANB Articaine and SUP Articaine - 2nd Molar | IANB Articaine and SUP Lidocaine - 1st Molar | IANB Articaine and SUP Lidocaine - 2nd Molar
Started | 28 | 24 | 36 | 40 | 35 | 38
Completed | 27 | 23 | 36 | 40 | 35 | 38
Not Completed | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Inadequate lip numbness: "missed" block | 1 | 1 | 0 | 0 | 0 | 0
Period: Supplemental Buccal Infiltration
Arm/Group | IANB Articaine Only - 1st Molar | IANB Articaine Only - 2nd Molar | IANB Articaine and SUP Articaine - 1st Molar | IANB Articaine and SUP Articaine - 2nd Molar | IANB Articaine and SUP Lidocaine - 1st Molar | IANB Articaine and SUP Lidocaine - 2nd Molar
Started (Supplemental buccal anesthesia (SUP) was provided in cases of unsuccessful IANB.) | 0 (No participants with successful IANB initially were brought forward to supplemental anesthetic) | 0 (No participants with successful IANB initially were brought forward to supplemental anesthetic) | 36 (Only after unsuccessful IANB.) | 40 (Only after unsuccessful IANB.) | 35 (Only after unsuccessful IANB.) | 38 (Only after unsuccessful IANB.)
Completed | 0 | 0 | 36 | 40 | 35 | 38
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall number of participants include all enrolled subjects that received the initial IANB anesthesia.
Groups:
- Total: Total of all reporting groups
Arm/Group | IANB Articaine Only - 1st Molar | IANB Articaine Only - 2nd Molar | IANB Articaine and SUP Articaine - 1st Molar | IANB Articaine and SUP Articaine - 2nd Molar | IANB Articaine and SUP Lidocaine - 1st Molar | IANB Articaine and SUP Lidocaine - 2nd Molar | Total
Number analyzed (Participants) | 28 | 24 | 36 | 40 | 35 | 38 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two subjects (1 first molar, 1 second molar) were excluded from analysis due to inadequate lip numbness ("missed block") after initial IANB Articaine.
  years
    number analyzed (Participants) | 27 | 23 | 36 | 40 | 35 | 38 | 199
    (all) | 35 (11) | 50 (18) | 40 (14) | 38 (15) | 35 (14) | 40 (14) | 39 (15)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two subjects (1 first molar, 1 second molar) were excluded from analysis due to inadequate lip numbness ("missed block") after initial IANB Articaine.
  Participants
    number analyzed (Participants) | 27 | 23 | 36 | 40 | 35 | 38 | 199
    Female | 13 | 13 | 12 | 23 | 22 | 19 | 102
    Male | 14 | 10 | 24 | 17 | 13 | 19 | 97
Region of Enrollment [Number; unit: participants] — Population: Two subjects (1 first molar, 1 second molar) were excluded from analysis due to inadequate lip numbness ("missed block") after initial IANB Articaine.
  participants
    United States: number analyzed (Participants) | 27 | 23 | 36 | 40 | 35 | 38 | 199
    United States | 27 | 24 | 36 | 40 | 35 | 38 | 199

OUTCOME MEASURES:

1. Primary Outcome: Anesthetic Success Rate of Supplemental Infiltration Injection
Description: Following an unsuccessful IANB, supplemental infiltration anesthesia with either articaine or lidocaine was given to achieve complete pulpal anesthesia
Time Frame: 5 min after injection
Measure: Count of Participants; unit: Participants
Groups:
- IANB Articaine and SUP Articaine - 1st Molar: Supplemental buccal anesthesia with articaine local anesthetic provided to 1st Molar after unsuccessful IANB.
- IANB Articaine and SUP Articaine - 2nd Molar: Supplemental buccal anesthesia with articaine local anesthetic provided to 2nd Molar after unsuccessful IANB.
- IANB Articaine and SUP Lidocaine - 1st Molar: Supplemental buccal anesthesia with lidocaine local anesthetic provided to 1st Molar after unsuccessful IANB.
- IANB Articaine and SUP Lidocaine - 2nd Molar: Supplemental buccal anesthesia with lidocaine local anesthetic provided to 2nd Molar after unsuccessful IANB.
Arm/Group | IANB Articaine and SUP Articaine - 1st Molar | IANB Articaine and SUP Articaine - 2nd Molar | IANB Articaine and SUP Lidocaine - 1st Molar | IANB Articaine and SUP Lidocaine - 2nd Molar
Number analyzed (Participants) | 36 | 40 | 35 | 38
Participants | 22 | 25 | 23 | 12
Statistical Analysis 1: Comparison: IANB Articaine and SUP Articaine - 1st Molar vs IANB Articaine and SUP Articaine - 2nd Molar; Test type: Superiority; p = .901, Chi-squared; We used the Chi-Square Test or Fisher's Exact test on the raw data depending on the number of data points in the table cells
Statistical Analysis 2: Comparison: IANB Articaine and SUP Lidocaine - 1st Molar vs IANB Articaine and SUP Lidocaine - 2nd Molar; Test type: Superiority; p = .004, Chi-squared; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Anesthetic Success Rate of an IANB With Articaine
Description: Success rate of an IANB with articaine using a conventional IANB technique
Time Frame: 15 min after injection
Population: All enrolled participants (N=201) received an IANB with Articaine. Two participants were excluded from data analysis due to inadequate lip numbness (IANB was considered "missed block"); thus N=199 were analyzed for success rate.
Measure: Count of Participants; unit: Participants
Groups:
- IANB Articaine - 1st Molar: Initial IANB (1.7cc 4% articaine with 1:100,000 epinephrine) provided to 1st Molar.
- IANB Articaine - 2nd Molar: Initial IANB (1.7cc 4% articaine with 1:100,000 epinephrine) provided to 2nd Molar.
Arm/Group | IANB Articaine - 1st Molar | IANB Articaine - 2nd Molar
Number analyzed (Participants) | 98 | 101
Participants | 27 | 23
Statistical Analysis 1: Comparison: IANB Articaine - 1st Molar vs IANB Articaine - 2nd Molar; Test type: Superiority; p = .437, Chi-squared; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Initial IANB Articaine: Initial IANB with articaine local anesthetic.
- SUP Articaine: Supplemental buccal anesthesia with articaine local anesthetic.
- SUP Lidocaine: Supplemental buccal anesthesia with lidocaine local anesthetic.
Arm/Group | Initial IANB Articaine | SUP Articaine | SUP Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/76 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/201 | 0/76 | 0/73
Other Adverse Events (participants affected / at risk) | 0/201 | 0/76 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes